CLINICAL TRIAL: NCT04203979
Title: Sepsis: From Syndrome to Personalized Care
Status: Recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Aleksander Rygh Holten, Principal Investigator, Oslo University Hospital
Other Study IDs: Sepsis-OUH-2
Record Dates: First submitted 2019-12-10; First posted 2019-12-18 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Sepsis Syndrome; Sepsis; Sepsis, Severe; Septic Shock
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Samples will be collected, together with routine blood samples, from patients with suspected sepsis shortly after arrival at the Emergency department, before antibiotics are given. Calprotectin, CRP and leukocytes wil be analysed in the routine laboratory. Blood will be biobanked for other analyses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective, observational study designed to examine the performance of biomarkers, molecular biological methods and other analysis in blood from patient with suspected sepsis in the Emergency department, as well as identidying novel sepsis endotypes. Around 1500 patients will be enrolled.

DETAILED DESCRIPTION:
The study will prospectively include adult patients (>18 years) with suspected sepsis admitted to Oslo University Hospital, Ullevål (OUH-Ullevål). Patients admitted to the emergency department and managed by the medical rapid response team or the sepsis rapid response team are considered eligible for inclusion. Informed consent will be collected at the emergency department if possible, or within few days, by a clinical investigator or a study nurse. The investigators aim to include 1500 patients treated by the Sepsis Rapid Response Team or Medical Emergency team for possible sepsis. Patients classified to have had other conditions than sepsis in the post hoc assessment will be used as controls. The inclusion period will be 3 years.

ELIGIBILITY:
Inclusion Criteria:

* admitted to emergency department OUH, Ullevål.
* managed by the medical rapid response team or the sepsis rapid response team

Exclusion Criteria:

* Not given informed consent by patient or next of kin (if patient is not able to)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with suspected sepsis or other severe conditions in the Emergency department.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2020-01-06 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of sepsis patient with elevated plasma-calprotectin | One year
  Sensitivity of plasma-calprotectin for detecting infections in critical ill medical patients in the Emergency department.
Area under the curve receiver operator characteristic (AUC - ROC) for inflammation biomarkers for detecting infection in critically ill patients. | One year
  Comparing area under the curve receiver operator characteristic (AUC - ROC) for calprotectin, pro-calcitonin, CRP and other biomarkers for detecting infections in critically ill patients in the Emergency department.
Number of sepsis patient with bacterial DNA detected in blood by molecular biological tests. | One year
  The performance of rapid molecular biological tests for detecting bacterial DNA in full blood in critically ill medical patients, compared to current state-of-the art diagnostics (blood culture).

SECONDARY OUTCOMES:
Concentration of biomarkers in blood. | One year
  Explore how the concentration of biomarkers of inflammation change during the course of the disease.

OTHER OUTCOMES:
Sepsis endotypes | 3 years
  Comprehensively characterize the host response to infection in patients presenting to the ED with sepsis and identify endotypes by unsupervised machine learning methods
Exteranal validation of sepsis endotypes | 3 years
  Externally validate host response profiles and multi-omic sepsis endotypes in two international cohorts.
Temperal profile of host response | 3 years
  Describe how host response profiles develop in the days after hospital admission and initiation of treatment.
E. coli influences the host respons | 3 years
  Characterize how genetic variation within E. coli influences the host response to sepsis

CONTACTS AND LOCATIONS:
Overall Officials: Aleksander R Holten, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Christensen EE, Binde C, Leegaard M, Tonby K, Dyrhol-Riise AM, Kvale D, Amundsen EK, Holten AR. DIAGNOSTIC ACCURACY AND ADDED VALUE OF INFECTION BIOMARKERS IN PATIENTS WITH POSSIBLE SEPSIS IN THE EMERGENCY DEPARTMENT. Shock. 2022 Oct 1;58(4):251-259. doi: 10.1097/SHK.0000000000001981. Epub 2022 Sep 6. PMID 36130401